CLINICAL TRIAL: NCT01030003
Title: The Impact of Sleep-Disordered Breathing on Adverse Pregnancy Outcomes
Brief Title: Snoring in Pregnancy and Adverse Maternal and Fetal Outcomes
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Louise O'Brien, Associate Professor, University of Michigan
Other Study IDs: R000038; 1R21HL089918-01A1 (NIH)
Record Dates: First submitted 2009-12-08; First posted 2009-12-10 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Sleep Apnea Syndromes
Keywords: Sleep-Disordered Breathing; Snoring; Pregnancy; Fetal Growth Retardation; Pre-Eclampsia
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring; Fetal Growth Retardation; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine the prevalence of sleep-disordered breathing in pregnant women during the third trimester of pregnancy and to investigate whether this is associated with high blood pressure in the mother and/or growth retardation in the baby.

ELIGIBILITY:
Inclusion Criteria:

* Women attending obstetric clinics at University of Michigan Hospitals.
* Willing and able to provide informed consent.
* Aged 18 years or older

Exclusion Criteria:

* Aged under 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible pregnant women are those receiving prenatal care and planning on delivering at the University of Michigan.
Sampling Method: Non-Probability Sample
Enrollment: 1685 (Actual)
Dates: Start 2007-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Maternal diagnosis of hypertension | 0-3 months after enrollment.

SECONDARY OUTCOMES:
Infant birth centile | 0-3 months after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Louise M O'Brien, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] O'Brien LM, Bullough AS, Owusu JT, Tremblay KA, Brincat CA, Chames MC, Kalbfleisch JD, Chervin RD. Snoring during pregnancy and delivery outcomes: a cohort study. Sleep. 2013 Nov 1;36(11):1625-32. doi: 10.5665/sleep.3112. PMID 24179294